CLINICAL TRIAL: NCT02113852
Title: Study of Blood, Tumor and Adjacent Normal Tissue Samples From Chinese Smoking Induced Lung Cancer Patients
Acronym: CHOICE
Status: Completed | Type: Observational
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CTONG 1308
Record Dates: First submitted 2014-03-24; First posted 2014-04-15 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non small cell Lung Cancer; Heavy smokers; Treatment naive patients
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — blood,tumor and adjacent normal tissue samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is an epidemiological,multicenter study of genomic and expression profiles of patients with newly diagnosed NSCLC.Two hundred and fifty NSCLC patients who fulfill the criteria are to be recruited by investigational sites.Approximately 100 of them will be from retrospectively collected samples with detailed clinical and 2-year follow-up information after surgeries.The demographics,cancer/adjacent normal tissue and matched blood sample will be collected after the patient had provided informed consent.All tissue samples will be analyzed for somatic mutations by exome deep sequencing,mRNA expression profiling by RNA sequencing and chromosome copy number variation by SNP array at the designated laboratories.

DETAILED DESCRIPTION:
The 2-year follow-up information of all enrolled patients will be collected every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent.
2. Male or female aged≥18 years.
3. .Histological or cytologically confirmed primary NSCLC，including histological subtypes:adenocarcinoma,squamous cell carcinoma and large cell carcinoma etc.
4. .Provision of surgical specimen and blood sample.The retrospective samples will be collected between 2006and 2012 from the bio-bank.
5. Patients must be willing to provide detailed clinical information (sex,age,geographic place,tumor stage,grade,size,smoking history,treatment history if any and outcome data).
6. Heavy smokers(defined as having smoked 20 pack-years or more).
7. Treatment naive patients:No prior chemotherapy,biological,immunological therapy or radical radiotherapy is permitted.

Exclusion Criteria:

* Not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study aims to collect approximately 250 smoking induced lung cancer(NSCLC) samples.Approximately 200 cases of treatment naive samples will be required. Samples will be collected mainly from the investigational sites in Guangzhou, Shanghai and Beijing that have expertise in lung cancer diagnosis.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-08; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
whole genome copy number variation in NSCLC patients | 2 years
  To indentify and characterize somatic mutations in coding region (exome) in NSCLC patients through next generation sequencing of the tumor and blood samples.To identify and characterize whole genome copy number variation in NSCLC patients by using the standard SNP array(Affymetrix SNP 6.0).To indentify and characterize the transcriptome of tumor versus adjacent normal tissues by using RNA sequencing.

SECONDARY OUTCOMES:
Establish more effective therapy for lung cancer treatment in the future | 2 years
  To identify the changes in molecular pathways and biomarker related to smoking induced lung cancer to help establish more effective therapy for lung cancer treatment in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Long Wu, MD, Principal Investigator — Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences